CLINICAL TRIAL: NCT01658150
Title: A Molecular Approach to Treat Cognition in Schizophrenia: Ca2+ Channel Blockade
Brief Title: Evaluating Isradipine for Cognitive Enhancement in Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Katherine Burdick, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 12-0679; HSM# 12-00311
Record Dates: First submitted 2012-07-12; First posted 2012-08-06 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognition; Schizophrenia; Schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Isradipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- isradipine (Experimental): open label
  Interventions: Drug: isradipine

INTERVENTIONS:
Drug: isradipine — Isradipine is a medication that acts by blocking a specific type of receptor in the brain called a calcium channel
  Other Names: Dynacirc CR

SUMMARY:
The purpose of this study is to evaluate the use of the drug isradipine for cognitive enhancement in patients diagnosed with schizophrenia and schizoaffective disorder.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of the drug isradipine for cognitive enhancement in patients diagnosed with schizophrenia and schizoaffective disorder. Incomplete treatment response can be common in these disorders. While there are medications that are effective at treating positive symptoms, some other symptoms of the disorders are often left only partially treated (cognitive impairment and negative symptoms). This study will begin to address if the medication isradipine might help to treat some of the cognitive problems associated with schizophrenia and schizoaffective disorder. Isradipine is a medication that acts by blocking a specific type of receptor in the brain called a calcium channel. It is currently approved by the FDA for hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* DSM-IV schizophrenia or schizoaffective disorder diagnosis
* Residual phase of illness criteria met at screen and baseline as defined by item scores of equal to or less than 4 on each of the Brief Psychiatric Rating Scale (BPRS) hallucinatory behavior, unusual thought content, conceptual disorganization items
* Hamilton Rating Scale for Depression (HRSD) equal to or less than 12
* Baseline Clinician Administered Scale for Mania (CARS-M) score of less than 5
* Simpson Angus Scale (SAS) total score equal to or less than 6
* Treatment with at least one but no more than two stably-dosed second-generation antipsychotic medication (other than clozapine) for equal to or greater than 2 months and no changes planned over the 4-week study period

Exclusion Criteria:

* History of CNS trauma, neurological disorder, ADHD, mental retardation, learning disability, or other non-schizophrenic cause of cognitive impairment
* DSM-IV diagnosis of substance abuse/dependence within 3 months
* Pregnant women or women of childbearing age who are not using a medically accepted means of contraception
* Women who are breastfeeding
* Active, unstable medical problem that may interfere with cognition
* Current treatment for hypertension
* Uncontrolled hypertension
* Any drug known to interact with isradipine
* History of GI strictures
* History of heart disease
* Abnormal lab or ECG at screen
* Significant suicidal ideation at baseline (HRSD item 3>2)
* ECT treatment within 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09; Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Burdick, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Isradipine: Isradipine is a medication that acts by blocking a specific type of receptor in the brain called a calcium channel. isradipine as utilized in this trial will be administered twice daily. Isradipine will be titrated as follows: baseline (week 0) 5 mg/day BID; Week 2 increase to 10 mg/day BID if 5 mg was well-tolerated. Dosing will be flexible based on side effects with a maximum=10 mg/day. If 5 mg cannot be tolerated, the subject will be discontinued.
Period: Overall Study
Arm/Group | Isradipine
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Isradipine
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: MATRICS Consensus Cognitive Battery (MCCB) Change in Neurocognitive/Functional Measures
Description: MATRICS Consensus Cognitive Battery (MCCB) as measure of Neurocognitive/Functional Measures is a standardized battery designed to measure cognitive functioning in people with schizophrenia. The MCCB is represented as a composite T score. A t score is a type of standard score computed by multiplying a z-score (how many standard deviations an element is from the mean) by 10 and adding 50.
Time Frame: baseline and week 4
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Isradipine
Number analyzed (Participants) | 10
z-score
  Baseline | 39.8 (13.2)
  Week 4 | 38.2 (12.6)

2. Primary Outcome: UPSA Communication Score
Description: UCSD Performance Skills Assessment (UPSA) - The UPSA is performance-based measure of real-world daily functioning abilities. Participants receive scores for the communication subscale (range = 0-20), with higher score indicating better neurocognitive functioning
Time Frame: baseline and week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale
  baseline | 15.3 (2.8)
  week 4 | 16.5 (2.0)

3. Primary Outcome: Quality of Life (QoL) Scale
Description: The QoL is a measure of the perceived satisfaction in an individual's daily life. This 16-item self-report measure is rated on a 7-point scale, ranging from 1 (terrible) to 7 (delighted), with a total score range from 16-112, where higher scores indicate higher satisfaction with daily life.
Time Frame: baseline and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale
  Baseline | 96.5 (15.5)
  Week 4 | 93.0 (16.9)

4. Secondary Outcome: Mean Change in PRISE Adverse Event Checklist Score
Description: The PRISE is a physician-administered checklist of adverse events. PRISE contains 33 items, each defined by an adverse event. Each item is rated on a 3-point scale, ranging from 0 (not present) to 2 (distressing), with a total score range from 0-66, where higher scores indicate more adverse events. Mean change for adverse events at week 4 as compared to baseline
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | -0.7 (2.7)

5. Secondary Outcome: Number of Participants With Normal ECG
Description: Number of participants with normal ECG readings to confirm inclusion into study and compared at week 4 to baseline
Time Frame: baseline and week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Isradipine
Number analyzed (Participants) | 10
Participants
  Baseline | 10
  Week 4 | 10

6. Secondary Outcome: Number of Participants With Normal Chemistry Panel
Description: Number of participants with normal chemistry panel to confirm inclusion into study at baseline and week
Time Frame: baseline and week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Isradipine
Number analyzed (Participants) | 10
Participants
  Baseline | 10
  Week 4 | 10

7. Secondary Outcome: Number of Participants With Normal Complete Blood Count (CBC)
Description: Number of participants with normal CBC to confirm inclusion into study at baseline and week 4
Time Frame: baseline and week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Isradipine
Number analyzed (Participants) | 10
Participants
  Baseline | 10
  Week 4 | 10

8. Secondary Outcome: Abnormal Involuntary Movement Scale (AIMS)
Description: Mean change for abnormal involuntary movements throughout the study. The AIMS is a physician-administered scale of abnormal involuntary movements. AIMS consists of 10 items, each defined by a series of movements. Each item is rated on a 5-point scale, ranging from 0 (not observed) to 4 (severe), with a total score range from 0-40, where higher scores indicate abnormal involuntary movements.
Time Frame: baseline and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | 0.7 (2.9)

9. Secondary Outcome: Modified Simpson Angus Scale (MSAS)
Description: Mean change for drug-induced disordered movement throughout the study. The MSAS is a physician-administered scale of abnormal drug-induced movements. MSAS consists of 6 items, each defined by a series of movements. Each item is rated on a 5-point scale, ranging form 0 (not observed) to 4 (most severe), with a total range of 0-24, where higher scores indicate drug-induced disordered movement.
Time Frame: baseline and week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | -0.3 (0.5)

10. Secondary Outcome: Beck Scale for Suicidal Ideation (SSI)
Description: a 21-question multiple choice, self-report inventory that is used for measuring the severity of suicidal ideation. Scoring is from a 0 (not at all) to 3 (severe) with a total score range of 0-63. Higher total scores indicate more severe suicidal ideation symptoms.
Time Frame: up to 4 weeks
Population: Data not collected.
Arm/Group | Isradipine
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Suicidal Acknowledgments
Description: Number of participants with Suicidal acknowledgements based on the Columbia Suicide Severity Rating Scales (C-SSRS) - Full range from 0 (low intensity suicidal ideation to 9 (high intensity suicidal ideation).
Time Frame: up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Isradipine
Number analyzed (Participants) | 10
Participants | 0

12. Secondary Outcome: Number of Participants With a Confirmed SCID-IV
Description: Number of participants with confirm diagnosis for inclusion into study using the Structured Clinical Interview for the DSM-IV (SCID-IV)
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Isradipine
Number analyzed (Participants) | 10
Participants | 10

13. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: Mean change for positive symptoms throughout the study. BPRS consists of 18 items, each defined by a series of symptoms. Each item is rated on a 7-point scale, ranging from 1 (not observed) to 7 (very severe), with a total score range from 18-126, where higher scores indicate psychiatric symptoms.
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | -1.0 (2.5)

14. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS)
Description: Mean change of negative symptoms throughout the study. SANS consists of 22 items, each defined by a series of symptoms. Each item is rated on a 6-point scale, ranging from 0 (no presence) to 5 (severe presence), with a total range of 0-110, where higher scores indicate negative symptoms.
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | -1.6 (3.3)

15. Secondary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: Mean change of symptoms of depression throughout the study. HRSD consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe), with a total score range of 0-56, where higher score indicates more depressive symptoms
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Isradipine: Isradipine is a medication that acts by blocking a specific type of receptor in the brain called a calcium channel. Need dosage information.
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | -0.6 (1.8)

16. Secondary Outcome: Clinical Global Impression Scale (CGI)
Description: Mean change of clinical impression of severity of psychiatric illness throughout the study. CGI consists of one item, defined by severity of illness. It is rated on a 7-point scale, ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients), with a total range score of 1-7, where higher score indicates severity of illness.
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | -0.2 (0.4)

17. Secondary Outcome: Clinician Administered Rating Scale for Mania (CARS-M)
Description: Mean change of symptoms of mania throughout the study. CARS-M contains 14 items rated from 0 (absent) to 5 (present) and one item scored 0 to 4, with total range from 0 to 74, where higher score indicates manic symptoms.
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isradipine
Number analyzed (Participants) | 10
score on a scale | 0 (0.7)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Isradipine
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Isradipine (N=11)
Nausea (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Poor coordination (General disorders) | 1
Blurred vision (Eye disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Frequent urination (Renal and urinary disorders) | 3
Menstrual irregular (Reproductive system and breast disorders) | 6
Difficulty sleeping (General disorders) | 4
Hypersomnia (General disorders) | 1
Loss of libido (Reproductive system and breast disorders) | 1
Anxiety (Psychiatric disorders) | 4
Poor concentration (General disorders) | 3
Restlessness (General disorders) | 2
Fatigue (General disorders) | 3
Decreased energy (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT01658150/Prot_SAP_000.pdf